CLINICAL TRIAL: NCT01074008
Title: A Blinded, Randomized, Placebo-controlled, Dose Ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Multiple Doses of ABT-450 With Ritonavir (ABT-450/r), ABT-333 or ABT-072 Each Administered Alone and in Combination With Peginterferon α-2a and Ribavirin (PegIFN/RBV) in Treatment-Naïve Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Randomized Study to Evaluate the Safety, Tolerability and Antiviral Activity of ABT-450, ABT-333 and ABT-072
Acronym: Champion2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M11-602
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis C; HCV; Chronic Hepatitis C Infection; Hepatitis C Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; ABT-072; dasabuvir; Ritonavir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- ABT-450/r (50/100 mg) once daily (QD) + pegIFN/RBV (Experimental): Participants received 50 mg ABT-450 and 100 mg ritonavir (r) monotherapy once daily for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-450; Drug: Ritonavir; Drug: Peginterferon alpha-2a; Drug: Ribavirin
- ABT-450/r (100/100 mg) once daily (QD) + pegIFN/RBV (Experimental): Participants received 100 mg ABT-450 and 100 mg ritonavir (r) monotherapy once daily for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-450; Drug: Ritonavir; Drug: Peginterferon alpha-2a; Drug: Ribavirin
- ABT-450/r (200/100 mg) once daily (QD) + pegIFN/RBV (Experimental): Participants received 200 mg ABT-450 and 100 mg ritonavir (r) monotherapy once daily for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-450; Drug: Ritonavir; Drug: Peginterferon alpha-2a; Drug: Ribavirin
- ABT-072 (100 mg) once daily (QD) + pegIFN/RBV (Experimental): Participants received 100 mg ABT-072 monotherapy once daily for 3 days followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-072; Drug: Peginterferon alpha-2a; Drug: Ribavirin
- ABT-072 (300 mg) once daily (QD) + pegIFN/RBV (Experimental): Participants received 300 mg ABT-072 monotherapy once daily for 3 days followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-072; Drug: Peginterferon alpha-2a; Drug: Ribavirin
- ABT-072 (600 mg) once daily (QD) + pegIFN/RBV (Experimental): Participants received 600 mg ABT-072 monotherapy once daily for 3 days followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-072; Drug: Peginterferon alpha-2a; Drug: Ribavirin
- ABT-333 (400 mg) twice a day (BID) + pegIFN/RBV (Experimental): Participants received 400 mg ABT-333 monotherapy twice a day for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-333; Drug: Peginterferon alpha-2a; Drug: Ribavirin
- ABT-333 (800 mg) twice daily (BID) + pegIFN/RBV (Experimental): Participants received 800 mg ABT-333 monotherapy twice a day for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: ABT-333; Drug: Peginterferon alpha-2a; Drug: Ribavirin
- Placebo + pegIFN/RBV (Placebo Comparator): Participants received matching placebo for ABT-450/r, ABT-072, or ABT-333 monotherapy at each dose level for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
  Interventions: Drug: Peginterferon alpha-2a; Drug: Ribavirin; Other: Placebo

INTERVENTIONS:
Drug: ABT-450 — 50 mg capsules co-administered with ritonavir
  Arms: ABT-450/r (100/100 mg) once daily (QD) + pegIFN/RBV; ABT-450/r (200/100 mg) once daily (QD) + pegIFN/RBV; ABT-450/r (50/100 mg) once daily (QD) + pegIFN/RBV
Drug: ABT-072 — 50 mg tablet
  Arms: ABT-072 (100 mg) once daily (QD) + pegIFN/RBV; ABT-072 (300 mg) once daily (QD) + pegIFN/RBV; ABT-072 (600 mg) once daily (QD) + pegIFN/RBV
Drug: ABT-333 — 400 mg tablet
  Other Names: Dasabuvir
  Arms: ABT-333 (400 mg) twice a day (BID) + pegIFN/RBV; ABT-333 (800 mg) twice daily (BID) + pegIFN/RBV
Drug: Ritonavir — 100 mg capsules co-administered with ABT-450
  Other Names: ABT-538; Norvir
  Arms: ABT-450/r (100/100 mg) once daily (QD) + pegIFN/RBV; ABT-450/r (200/100 mg) once daily (QD) + pegIFN/RBV; ABT-450/r (50/100 mg) once daily (QD) + pegIFN/RBV
Drug: Peginterferon alpha-2a — Syringe, 180 µg/0.5 mL for subcutaneous injections
Drug: Ribavirin — 200 mg tablet dosed at 1000 or 1200 mg daily divided twice a day
Other: Placebo — Matching placebo for ABT-450/r, ABT-072, or ABT-333 monotherapy at each dose level
  Arms: Placebo + pegIFN/RBV

SUMMARY:
This study assessed the safety, tolerability, pharmacokinetics, and antiviral activity of multiple oral doses of ABT-450/ritonavir (r), ABT-333 (also known as dasabuvir), or ABT-072 in hepatitis C virus (HCV), genotype 1-infected, treatment-naïve adults.

DETAILED DESCRIPTION:
This was a Phase 2a, randomized, blinded, placebo-controlled, dose-ranging study in chronically, hepatitis C virus (HCV) genotype 1-infected participants designed to explore the safety, tolerability, pharmacokinetics, antiviral activity, as well as the evolution and persistence to resistance of ABT-450/r, ABT-333, or ABT-072. Participants were treated with ABT-450/r, ABT-333, or ABT-072 monotherapy for 3 days, followed by 81 days (12 weeks minus 3 days of monotherapy) of ABT-450/r, ABT-333, or ABT-072 combined with pegylated interferon/ribavirin (pegIFN/RBV), followed by 36 weeks of pegIFN/RBV alone. Participants randomized to an ABT-450/r treatment group who achieved rapid virologic response (RVR) and had HCV ribonucleic acid (RNA) levels < 25 IU/mL at all subsequent visits were eligible to stop pegIFN/RBV therapy on or after Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C virus (HCV), genotype 1 infection (HCV ribonucleic acid level greater than or equal to 100,000 IU/mL) at screening
* Liver biopsy within 3 years with histology consistent with HCV-induced liver damage, with no evidence of cirrhosis or liver pathology due to any cause other than chronic HCV
* Treatment naïve male or female between the ages of 18 and 65
* Females must be post-menopausal for more than 2 years or surgically sterile
* Negative screen for drugs and alcohol
* Negative hepatitis B surface antigen (HBsAg) and anti-human immunodeficiency virus antibodies (anti-HIV Ab)
* No use of cytochrome P450 3A (CYP3A) and cytochrome P450 2C8 (CYP2C8) enzyme inducers or inhibitors within 1 month of dosing
* Be in a condition of general good health, as perceived by the investigator, other than HCV infection

Exclusion Criteria:

* Significant sensitivity to any drug
* Use of herbal supplements within 2 weeks prior to study drug dosing
* History of major depression within 2 years
* Prior treatment with any investigational or commercially available anti-HCV agents
* Abnormal laboratory tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, Study Director — AbbVie
Locations (26):
- United States (25):
  - Site Reference ID/Investigator# 23392, Phoenix, Arizona
  - Site Reference ID/Investigator# 23370, Anaheim, California
  - Site Reference ID/Investigator# 23387, La Jolla, California
  - Site Reference ID/Investigator# 23388, Los Angeles, California
  - Site Reference ID/Investigator# 23371, Aurora, Colorado
  - Site Reference ID/Investigator# 23369, Orlando, Florida
  - Site Reference ID/Investigator# 26362, Orlando, Florida
  - Site Reference ID/Investigator# 23373, Chicago, Illinois
  - Site Reference ID/Investigator# 24908, Chicago, Illinois
  - Site Reference ID/Investigator# 23381, Indianapolis, Indiana
  - Site Reference ID/Investigator# 23372, Baton Rouge, Louisiana
  - Site Reference ID/Investigator# 24710, New Orleans, Louisiana
  - Site Reference ID/Investigator# 23391, Baltimore, Maryland
  - Site Reference ID/Investigator# 23377, Detroit, Michigan
  - Site Reference ID/Investigator# 24909, Saint Paul, Minnesota
  - Site Reference ID/Investigator# 35842, New York, New York
  - Site Reference ID/Investigator# 23379, New York, New York
  - Site Reference ID/Investigator# 23375, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 23385, Durham, North Carolina
  - Site Reference ID/Investigator# 23376, Dallas, Texas
  - Site Reference ID/Investigator# 24891, Houston, Texas
  - Site Reference ID/Investigator# 23382, San Antonio, Texas
  - Site Reference ID/Investigator# 24715, Salt Lake City, Utah
  - Site Reference ID/Investigator# 25463, Seattle, Washington
  - Site Reference ID/Investigator# 23383, Madison, Wisconsin
- Site Reference ID/Investigator# 23363, Ponce, Puerto Rico

REFERENCES:
- [Derived] Pilot-Matias T, Tripathi R, Cohen D, Gaultier I, Dekhtyar T, Lu L, Reisch T, Irvin M, Hopkins T, Pithawalla R, Middleton T, Ng T, McDaniel K, Or YS, Menon R, Kempf D, Molla A, Collins C. In vitro and in vivo antiviral activity and resistance profile of the hepatitis C virus NS3/4A protease inhibitor ABT-450. Antimicrob Agents Chemother. 2015 Feb;59(2):988-97. doi: 10.1128/AAC.04227-14. Epub 2014 Dec 1. PMID 25451053
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV | Placebo + pegIFN/RBV
Started | 8 | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 11
Completed Direct-acting Antiviral Agent | 8 | 7 | 7 | 8 | 8 | 5 | 8 | 7 | 5
Completed | 7 | 5 | 6 | 7 | 6 | 7 | 7 | 8 | 7
Not Completed | 1 | 3 | 2 | 1 | 2 | 0 | 1 | 0 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 4

BASELINE CHARACTERISTICS:
Population: All participants who recieved at least one dose of study drug were included in the baseline characteristic analaysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV | Placebo + pegIFN/RBV | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 11 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.36) | 50.9 (2.59) | 50.6 (9.26) | 53.5 (5.40) | 51.3 (7.76) | 40.9 (11.25) | 49.6 (8.37) | 53.5 (6.46) | 51.5 (6.36) | 50.2 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 3 | 1 | 0 | 2 | 0 | 2 | 16
  Male | 7 | 5 | 4 | 5 | 7 | 7 | 6 | 8 | 9 | 58

OUTCOME MEASURES:

1. Primary Outcome: Maximal Change From Baseline in Hepatitis C Virus Ribonucleic Acid (HCV RNA) Levels During ABT-450/r, ABT-333, or ABT-072 Monotherapy Treatment
Description: Plasma HCV RNA levels (reported as log10 IU/mL) were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay that had a lower limit of detection of 10 IU/mL and a lower limit of quantification of 25 IU/mL. The baseline value was the HCV RNA level before the first dose of study drug on Day 1. The maximal change during monotherapy was the difference from baseline to the lowest log10 HCV RNA level anytime after the first dose of study drug on Day 1 through the last log10 HCV RNA level before the first dose of study drug on Day 4. Data are reported as the mean ± standard deviation.
Time Frame: Prior to dosing on Day 1 to before the morning dose on Day 4
Population: Participants received at least one dose of study drug (direct-acting antiviral agent) and have both baseline and at least one post-baseline measurement of HCV RNA levels during monotherapy treatment.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 11
log10 IU/mL | -4.07 (0.53) | -3.91 (0.42) | -4.11 (0.32) | -1.14 (0.99) | -1.07 (0.41) | -1.57 (0.94) | -1.08 (0.68) | -0.95 (0.68) | -0.36 (0.13)
Statistical Analysis 1: Comparison: ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Eight participants per ABT-450/r group and 11 participants in the placebo group would provide > 95% power to detect a 1.0 log10 difference with a common standard deviation of 0.5 log10 IU/mL using a two-sided, two-sample t-test with a significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANCOVA — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05; Treatment was the factor and baseline log10 HCV RNA level was the covariate
Statistical Analysis 2: Comparison: ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05; Treatment was the factor and baseline log10 HCV RNA level was the covariate
Statistical Analysis 3: Comparison: ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05; Treatment was the factor and baseline log10 HCV RNA level was the covariate
Statistical Analysis 4: Comparison: ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Eight participants per ABT-072 and 11 participants in the placebo group would provide 92% power to detect a 1.0 log10 difference with a standard deviation of 0.6 log10 IU/mL and a two-sided, two-sample t-test with a significance level of 0.05; Test type: Superiority or Other; p = 0.009, ANCOVA — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05; Treatment was the factor and baseline log10 HCV RNA level was the covariate
Statistical Analysis 5: Comparison: ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.012, ANCOVA — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05; Treatment was the factor and baseline log10 HCV RNA level was the covariate
Statistical Analysis 6: Comparison: ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.001, ANCOVA — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05; Treatment was the factor and baseline log10 HCV RNA level was the covariate
Statistical Analysis 7: Comparison: ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Eight subjects per ABT-333 group and 11 subjects in the placebo group would provide 82% power to detect a 1.0 log10 IU/mL difference with a standard deviation of 0.7 log10 IU/mL and a 2-sided 2-sample t-test with a significance level of 0.05; Test type: Superiority or Other; p = 0.032, ANCOVA — There was no adjustment for multiple comparisons and the pre-specified, 2-sided significance level was ≤ 0.05; Treatment was the factor and baseline log10 HCV RNA level was the covariate
Statistical Analysis 8: Comparison: ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Eight participants per ABT-333 group and 11 participants in the placebo group would provide 82% power to detect a 1.0 log10 IU/mL difference with a standard deviation of 0.7 log10 IU/mL and a two-sided, two-sample t-test with a significance level of 0.05; Test type: Superiority or Other; p = 0.053, ANCOVA — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05; Treatment was the factor and baseline log10 HCV RNA level was the covariate

2. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR) at Week 4
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay that had a lower limit of detection of 10 IU/mL and a lower limit of quantification (LLOQ) of 25 IU/mL. Rapid virologic response was defined as HCV RNA level < LLOQ (< 25 IU/mL) at Week 4. Data are reported as the percentage of participants with RVR.
Time Frame: Week 4
Population: All participants who received at least one dose of study drug and had at least one post-baseline HCV RNA value were included in this efficacy analysis.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 11
percentage of participants | 87.5 | 75.0 | 100.0 | 37.5 | 12.5 | 42.9 | 50.0 | 50.0 | 9.1
Statistical Analysis 1: Comparison: ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.001, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 2: Comparison: ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.006, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 3: Comparison: ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p < 0.001, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 4: Comparison: ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.262, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 5: Comparison: ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 1.000, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 6: Comparison: ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.245, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 7: Comparison: ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.111, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 8: Comparison: ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.111, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05

3. Secondary Outcome: Percentage of Participants With Partial Early Virologic Response (EVR) at Week 12
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay that had a lower limit of detection of 10 IU/mL and a lower limit of quantification of 25 IU/mL. Partial early virologic response (EVR) was defined as HCV RNA levels that decreased > 2 log10 IU/mL at Week 12 as compared to baseline. The baseline value was the last measurement before the first dose on Day 1. Data are reported as the percentage of participants with partial EVR.
Time Frame: Baseline and Week 12
Population: To be included in the efficacy analysis, participants received at least one dose of study drug (direct-acting antiviral agent) and at least one post-baseline measurement of HCV RNA levels.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 11
percentage of participants | 100.0 | 87.5 | 100.0 | 100.0 | 62.5 | 100.0 | 100.0 | 100.0 | 36.4
Statistical Analysis 1: Comparison: ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.013, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 2: Comparison: ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.059, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 3: Comparison: ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.013, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 4: Comparison: ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.013, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 5: Comparison: ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.370, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 6: Comparison: ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.013, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 7: Comparison: ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.013, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 8: Comparison: ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.013, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of ABT-450
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-450 using validated analytical methods. The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that a drug achieves in the blood after administration in a dosing interval. The Cmax of ABT-450 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: Immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose)
Population: All participants who received at least one dose of study drug (direct-acting antiviral agent) were included in the pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 34.4 (31.7) | 165 (221) | 2923 (2026)

5. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of ABT-450
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-450 using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in hours) is the time it takes for a drug to achieve Cmax. The Tmax of ABT-450 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
Hours | 2.5 (0.9) | 4.8 (3.5) | 3.0 (1.1)

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24) Post-dose of ABT-450
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-450 using validated analytical methods. The area under the plasma concentration-time curve (AUC; measured in ng*hr/mL) is a method of measurement to determine the total exposure of a drug in blood plasma. The AUC24 of ABT-450 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL | 250 (245) | 1122 (992) | 17351 (15841)

7. Primary Outcome: Maximum Plasma Concentration (Cmax) of Ritonavir
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ritonavir using validated analytical methods. The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that a drug achieves in the blood after administration in a dosing interval. The Cmax of ritonavir was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 563 (674) | 851 (638) | 1098 (619)

8. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Ritonavir
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ritonavir using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in hours) is the time it takes for a drug to achieve Cmax. The Tmax of ritonavir was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
Hours | 4.8 (2.8) | 5.3 (3.2) | 4.5 (1.4)

9. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24) Post-dose of Ritonavir
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ritonavir using validated analytical methods. The area under the plasma concentration-time curve (AUC; measured in ng*hr/mL) is a method of measurement to determine the total exposure of a drug in blood plasma. The AUC24 of ritonavir was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
ng*hr/mL | 4518 (5063) | 7638 (6284) | 8663 (5006)

10. Primary Outcome: Maximum Plasma Concentration (Cmax) of ABT-072
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-072 using validated analytical methods. The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that a drug achieves in the blood after administration in a dosing interval. The Cmax of ABT-072 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 7
ng/mL | 390 (153) | 1218 (382) | 1748 (707)

11. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of ABT-072
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-072 using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in hours) is the time it takes for a drug to achieve Cmax. The Tmax of ABT-072 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 7
Hours | 4.5 (1.4) | 2.8 (1.0) | 3.1 (1.1)

12. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24) Post-dose of ABT-072
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-072 using validated analytical methods. The area under the plasma concentration-time curve (AUC; measured in ng*hr/mL) is a method of measurement to determine the total exposure of a drug in blood plasma. The AUC24 of ABT-072 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 7
ng*hr/mL | 3678 (1742) | 9413 (3125) | 14126 (6102)

13. Primary Outcome: Maximum Plasma Concentration (Cmax) of ABT-333
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-333 using validated analytical methods. The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that a drug achieves in the blood after administration in a dosing interval. The Cmax of ABT-333 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV
Number analyzed (Participants) | 8 | 6
ng/mL | 800 (382) | 1201 (419)

14. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of ABT-333
Description: Blood samples were collected immediately prior to morning dose (time 0 hours); 2, 4, 8, 12, and 16 hours after the morning dose on Day 1; and prior to dose on Day 2 (24 hours after Day 1 dose). The samples were analyzed for the concentration of ABT-333 using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in hours) is the time it takes for a drug to achieve Cmax. The Tmax of ABT-333 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV
Number analyzed (Participants) | 8 | 6
Hours | 4.5 (5.2) | 7.0 (8.4)

15. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 12 Hours (AUC12) Post-dose of ABT-333
Description: Blood samples were collected immediately prior to morning dose (time 0 hours) and at 2, 4, 8, and 12 hours after the morning dose on Day 1. The samples were analyzed for the concentration of ABT-333 using validated analytical methods. The area under the plasma concentration-time curve (AUC; measured in ng*hr/mL) is a method of measurement to determine the total exposure of a drug in blood plasma. The AUC12 of ABT-333 was estimated using non-compartmental methods and data are reported as the mean ± standard deviation.
Time Frame: Immediately prior to morning dose (time 0 hours) and at 2, 4, 8, and 12 hours after the morning dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV
Number analyzed (Participants) | 8 | 6
ng*hr/mL | 4315 (2176) | 6431 (1914)

16. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR) at Week 12
Description: Plasma hepatitis C virus ribonucleic acid (HCV RNA) levels were determined for each sample using a real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay that had a lower limit of detection of 10 IU/mL and a lower limit of quantification (LLOQ) of 25 IU/mL. Complete EVR was defined as HCV RNA levels < LLOQ (< 25 IU/mL) at Week 12. Data are reported as the percentage of participants with cEVR.
Time Frame: Week 12
Population: To be included in the efficacy analysis, participants received at least one dose of study drug (direct-acting antiviral agent) and have at least one post-baseline measurement of HCV RNA levels.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV | Placebo + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 11
percentage of participants | 87.5 | 87.5 | 100.0 | 75.0 | 50.0 | 85.7 | 87.5 | 62.5 | 18.2
Statistical Analysis 1: Comparison: ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.005, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 2: Comparison: ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.005, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 3: Comparison: ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p < 0.001, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 4: Comparison: ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.024, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 5: Comparison: ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.319, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 6: Comparison: ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.013, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 7: Comparison: ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.005, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05
Statistical Analysis 8: Comparison: ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV vs Placebo + pegIFN/RBV; Test type: Superiority or Other; p = 0.074, Fisher Exact — There was no adjustment for multiple comparisons and the pre-specified, two-sided significance level was ≤ 0.05

17. Other Pre Specified Outcome: Number of Participants With Resistance-Associated Variants and Phenotypic Resistance to ABT-450 in Non-structural Viral Protein 3 (NS3)
Description: Baseline samples were analyzed for resistance-associated amino acid variants using population and clonal sequencing and were compared with the appropriate reference sequence (1a-H77 or 1b-Con1). Phenotypic resistance to ABT-450 at baseline was assessed by calculating the fold difference in the half maximal effective concentration (EC50) compared with the EC50 for the appropriate reference replicon (1a-H77 or 1b-Con1). Available samples at Day 4 with HCV RNA ≥ 1000 IU/mL were analyzed for resistance-associated variants using population and clonal sequencing and were compared with the baseline sequences to assess amino acid changes. Phenotypic resistance to ABT-450 at Day 4 was assessed by calculating the fold difference in the EC50 compared with the EC50 for the corresponding baseline sample. The number of participants with variants at resistance-associated amino acid positions and phenotypic resistance are presented.
Time Frame: Baseline and Day 4
Population: All participants who received at least one dose of study drug (direct-acting antiviral agent) were included in the analysis. When the number of participants used to analyze the data at a specific time point differs from the Number of Participants Analyzed, the n (number of participants) is denoted in the Category Title.
Measure: Number; unit: participants
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (100/100 mg) Once Daily (QD) + pegIFN/RBV | ABT-450/r (200/100 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 8
participants
  Baseline Variants in NS3 | 0 | 0 | 0
  Baseline Resistance to ABT-450 >10-fold | 0 | 0 | 0
  Day 4 Variants in NS3 (n=3, 2, 3) | 2 | 2 | 1
  Day 4: Resistance to ABT-450 >10-fold (n=3, 2, 3) | 1 | 1 | 0

18. Other Pre Specified Outcome: Number of Participants With Resistance-Associated Variants and Phenotypic Resistance to ABT-072 in Non-structural Viral Protein 5B (NS5B)
Description: Baseline samples were analyzed for resistance-associated amino acid variants using population and clonal sequencing and were compared with the appropriate reference sequence (1a-H77 or 1b-Con1). Phenotypic resistance to ABT-072 at baseline was assessed by calculating the fold difference in the half maximal effective concentration (EC50) compared with the EC50 for the appropriate reference replicon (1a-H77 or 1b-Con1). Available samples at Day 4 with HCV RNA ≥ 1000 IU/mL were analyzed for the presence of resistance-associated variants using population and clonal sequencing and were compared with the baseline sequences to assess amino acid changes. Phenotypic resistance to ABT-072 at Day 4 was assessed by calculating the fold difference in the EC50 compared with the EC50 for the corresponding baseline sample. The number of participants with variants at resistance-associated amino acid positions and phenotypic resistance are presented.
Time Frame: Baseline and Day 4
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | ABT-072 (100 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (300 mg) Once Daily (QD) + pegIFN/RBV | ABT-072 (600 mg) Once Daily (QD) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8 | 7
participants
  Baseline Variants in NS5B | 0 | 1 | 0
  Baseline Resistance to ABT-072 >10-fold | 0 | 1 | 0
  Day 4: Variants in NS5B (n=6, 7, 6) | 1 | 2 | 1
  Day 4: Resistance to ABT-072 >10-fold (n=6, 7, 6) | 0 | 0 | 1

19. Other Pre Specified Outcome: Number of Participants With Resistance-Associated Variants and Phenotypic Resistance to ABT-333 in Non-structural Viral Protein 5B (NS5B)
Description: Baseline samples were analyzed for resistance-associated amino acid variants using population and clonal sequencing and were compared with the appropriate reference sequence (1a-H77 or 1b-Con1). Phenotypic resistance to ABT-333 at baseline was assessed by calculating the fold difference in the half maximal effective concentration (EC50) compared with the EC50 for the appropriate reference replicon (1a-H77 or 1b-Con1). Available samples at Day 4 with HCV RNA ≥ 1000 IU/mL were analyzed for the presence of resistance-associated variants using population and clonal sequencing and were compared with the baseline sequences to assess amino acid changes. Phenotypic resistance to ABT-333 at Day 4 was assessed by calculating the fold difference in the EC50 compared with the EC50 for the corresponding baseline sample. The number of participants with variants at resistance-associated amino acid positions and phenotypic resistance are presented.
Time Frame: Baseline and Day 4
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | ABT-333 (400 mg) Twice a Day (BID) + pegIFN/RBV | ABT-333 (800 mg) Twice Daily (BID) + pegIFN/RBV
Number analyzed (Participants) | 8 | 8
participants
  Baseline Variants in NS5B | 1 | 2
  Baseline Resistance to ABT-333 >10-fold NS5B | 0 | 1
  Day 4: Variants in NS5B (n=7, 8) | 3 | 3
  Day 4: Resistance to ABT-333 >10-fold (n=7, 8) | 0 | 0

20. Other Pre Specified Outcome: Change From Baseline in Hepatitis C Virus Patient-reported Outcomes (HCV-PRO) Total Score
Description: The Hepatitis C Virus Patient-report Outcomes (HCV-PRO, formerly known as HCV Quality of Life) survey was used to assess disease-specific function and well-being on a scale from 0 to 100; a higher score indicated relatively good function and well-being of treated participants. Data presented are the summaries across all participants, for each treatment arm, regardless of dose. Data are reported as the group mean change from baseline ± standard deviation.
Time Frame: Baseline up to Post-treatment Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ABT-450/r (Regardless of Dose) + pegIFN/RBV: Participants received ABT-450 and ritonavir (r) monotherapy at each dose level once daily for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 μg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-072 (Regardless of Dose) + pegIFN/RBV: Participants received ABT-072 monotherapy at each dose level once daily for 3 days followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 μg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-333 (Regardless of Dose) + pegIFN/RBV: Participants received ABT-333 monotherapy at each dose level twice a day for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 μg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- Placebo (Regardless of Dose) + pegIFN/RBV: Participants received matching placebo for ABT-450/r, ABT-072, or ABT-333 monotherapy at each dose level for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 μg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
Arm/Group | ABT-450/r (Regardless of Dose) + pegIFN/RBV | ABT-072 (Regardless of Dose) + pegIFN/RBV | ABT-333 (Regardless of Dose) + pegIFN/RBV | Placebo (Regardless of Dose) + pegIFN/RBV
Number analyzed (Participants) | 12 | 13 | 10 | 4
units on a scale | -0.78 (15.53) | -0.37 (13.97) | -3.25 (14.72) | -9.04 (12.41)

21. Other Pre Specified Outcome: Change From Baseline in ED-5D Visual Analog Scale (ED-5D VAS) Score
Description: The ED-5D VAS was a self-rating survey used to capture the current health status of a participant and ranged from 0 (the worst imaginable health state) to 100 (best imaginable health state). Data presented are the summaries across all participants, for each treatment arm, regardless of dose. Data are presented as the group mean change from baseline ± standard deviation.
Time Frame: Baseline and Post-treatment Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABT-450/r (Regardless of Dose) + pegIFN/RBV | ABT-072 (Regardless of Dose) + pegIFN/RBV | ABT-333 (Regardless of Dose) + pegIFN/RBV | Placebo (Regardless of Dose) + pegIFN/RBV
Number analyzed (Participants) | 11 | 13 | 11 | 4
units on a scale | -5.91 (31.92) | -2.38 (29.86) | 11.18 (27.19) | -9.00 (22.23)

22. Other Pre Specified Outcome: Change From Baseline in EQ-5D (3 Level) Health Index Score
Description: The EQ-5D was a health state questionnaire used to measure five health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The combination of responses from all five dimensions were derived into an index score ranging from 0 to 1; a higher score indicated a more preferable health utility value from the societal perspectives. Data presented are the summaries across all participants, for each treatment arm, regardless of dose. Data are presented as the group mean change from baseline ± standard deviation.
Time Frame: Baseline and Post-treatment Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABT-450/r (Regardless of Dose) + pegIFN/RBV | ABT-072 (Regardless of Dose) + pegIFN/RBV | ABT-333 (Regardless of Dose) + pegIFN/RBV | Placebo (Regardless of Dose) + pegIFN/RBV
Number analyzed (Participants) | 12 | 13 | 11 | 4
units on a scale | -0.06 (0.22) | -0.06 (0.15) | -0.02 (0.17) | -0.09 (0.09)

23. Other Pre Specified Outcome: Change From Baseline in SF-36 Physical Component Summary (PCS)
Description: The Physical Component Summary (PCS) of the SF-36 was used to measure the overall physical health status of a participant. The aggregated score of the SF-36 PCS score was standardized using a linear T-score transformation with a mean of 50 and a standard deviation of 10; a higher score indicated better physical function and well-being. Data presented are the summaries across all participants, for each treatment arm, regardless of dose. Data are presented as the group mean change from baseline ± standard deviation.
Time Frame: Baseline and Post-treatment Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABT-450/r (Regardless of Dose) + pegIFN/RBV | ABT-072 (Regardless of Dose) + pegIFN/RBV | ABT-333 (Regardless of Dose) + pegIFN/RBV | Placebo (Regardless of Dose) + pegIFN/RBV
Number analyzed (Participants) | 11 | 13 | 11 | 4
units on a scale | 3.01 (6.15) | -1.92 (5.89) | 4.08 (5.76) | -2.84 (7.92)

24. Other Pre Specified Outcome: Change From Baseline in SF-36 Mental Component Summary (MCS)
Description: The Mental Component Summary (MCS) of the SF-36 was used to measure the overall mental health status of participants. The aggregated score of the SF-36 MPS was standardized using a linear T-score transformation with a mean of 50 and a standard deviation of 10; a higher score indicated better mental function and well-being. Data presented are the summaries across all participants, for each treatment arm, regardless of dose. Data are presented as the group mean change from baseline ± standard deviation.
Time Frame: Baseline and Post-treatment Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABT-450/r (Regardless of Dose) + pegIFN/RBV | ABT-072 (Regardless of Dose) + pegIFN/RBV | ABT-333 (Regardless of Dose) + pegIFN/RBV | Placebo (Regardless of Dose) + pegIFN/RBV
Number analyzed (Participants) | 11 | 13 | 11 | 4
units on a scale | -2.77 (5.99) | -0.41 (10.64) | -4.37 (11.00) | -10.29 (11.35)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration to 30 days after last dose of ABT-450/r, ABT-267, or ABT-333 (16 Weeks); Serious adverse events were also collected from the time that informed consent was obtained (76 weeks ).
Groups:
- ABT-450/r (50/100 mg) Once Daily (QD) + (pegIFN/RBV): Participants received 50 mg ABT-450 and 100 mg ritonavir (r) monotherapy once daily for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-450/r (100/100 mg) Once Daily (QD) + (pegIFN/RBV): Participants received 100 mg ABT-450 and 100 mg ritonavir (r) monotherapy once daily for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-450/r (200/100 mg) Once Daily (QD) + (pegIFN/RBV): Participants received 200 mg ABT-450 and 100 mg ritonavir (r) monotherapy once daily for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-072 (100 mg) Once Daily (QD) + (pegIFN/RBV): Participants received 100 mg ABT-072 monotherapy once daily for 3 days followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-072 (300 mg) Once Daily (QD) + (pegIFN/RBV): Participants received 300 mg ABT-072 monotherapy once daily for 3 days followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-072 (600 mg) Once Daily (QD) + (pegIFN/RBV: Participants received 600 mg ABT-072 monotherapy once daily for 3 days followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-333 (400 mg) Twice a Day (BID) + (pegIFN/RBV): Participants received 400 mg ABT-333 monotherapy twice a day for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- ABT-333 (800 mg) Twice Daily (BID) + (pegIFN/RBV): Participants received 800 mg ABT-333 monotherapy twice a day for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
- Placebo + (pegIFN/RBV): Participants received matching placebo for ABT-450/r, ABT-072, or ABT-333 monotherapy at each dose level for 3 days, followed by the addition of pegylated interferon/ribavirin (pegIFN/RBV) for a total of 12 weeks of combination treatment, followed by 36 weeks of pegIFN/RBV alone. Pegylated interferon was dosed at 180 µg subcutaneously once a week and RBV was dosed 1000 or 1200 mg daily divided twice a day.
Arm/Group | ABT-450/r (50/100 mg) Once Daily (QD) + (pegIFN/RBV) | ABT-450/r (100/100 mg) Once Daily (QD) + (pegIFN/RBV) | ABT-450/r (200/100 mg) Once Daily (QD) + (pegIFN/RBV) | ABT-072 (100 mg) Once Daily (QD) + (pegIFN/RBV) | ABT-072 (300 mg) Once Daily (QD) + (pegIFN/RBV) | ABT-072 (600 mg) Once Daily (QD) + (pegIFN/RBV | ABT-333 (400 mg) Twice a Day (BID) + (pegIFN/RBV) | ABT-333 (800 mg) Twice Daily (BID) + (pegIFN/RBV) | Placebo + (pegIFN/RBV)
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/8 | 1/8 | 0/8 | 0/7 | 0/8 | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 8/8 | 8/8 | 7/7 | 8/8 | 8/8 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r (50/100 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-450/r (100/100 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-450/r (200/100 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-072 (100 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-072 (300 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-072 (600 mg) Once Daily (QD) + (pegIFN/RBV (N=7) | ABT-333 (400 mg) Twice a Day (BID) + (pegIFN/RBV) (N=8) | ABT-333 (800 mg) Twice Daily (BID) + (pegIFN/RBV) (N=8) | Placebo + (pegIFN/RBV) (N=11)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r (50/100 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-450/r (100/100 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-450/r (200/100 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-072 (100 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-072 (300 mg) Once Daily (QD) + (pegIFN/RBV) (N=8) | ABT-072 (600 mg) Once Daily (QD) + (pegIFN/RBV (N=7) | ABT-333 (400 mg) Twice a Day (BID) + (pegIFN/RBV) (N=8) | ABT-333 (800 mg) Twice Daily (BID) + (pegIFN/RBV) (N=8) | Placebo + (pegIFN/RBV) (N=11)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 2 | 1 | 2 | 2 | 0 | 2 | 2 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1 | 5 | 1 | 2 | 1 | 1 | 2 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MACULAR OEDEMA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RETINAL DETACHMENT (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
RETINAL EXUDATES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 2 | 2 | 2 | 3 | 4
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
DYSPEPSIA (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GINGIVITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GLOSSODYNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
LIP DRY (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
LOOSE TOOTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 2 | 2 | 1 | 3 | 4
PROCTALGIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROCTITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1
APPLICATION SITE RASH (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
CHILLS (General disorders) | 2 | 1 | 1 | 1 | 2 | 0 | 2 | 2 | 0
FATIGUE (General disorders) | 3 | 4 | 3 | 6 | 3 | 3 | 4 | 3 | 6
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 2 | 2 | 2 | 2 | 0 | 1 | 4 | 1
INFUSION SITE INFLAMMATION (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
INJECTION SITE HAEMATOMA (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INJECTION SITE RASH (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
INJECTION SITE REACTION (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
IRRITABILITY (General disorders) | 2 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 1
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PAIN (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0
PYREXIA (General disorders) | 3 | 1 | 1 | 2 | 2 | 0 | 2 | 1 | 1
TEMPERATURE INTOLERANCE (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
THIRST (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HEPATOMEGALY (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CANDIDIASIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
PERITONSILLAR ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 0 | 3 | 1 | 0 | 1
AXILLARY MASS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 4
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 2 | 1 | 3 | 0 | 1 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1
DIZZINESS (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 3 | 0 | 2 | 4
DYSGEUSIA (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 2
HEADACHE (Nervous system disorders) | 6 | 4 | 5 | 7 | 5 | 5 | 2 | 4 | 4
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
ABNORMAL DREAMS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
AFFECT LABILITY (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ANGER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 1 | 3 | 0 | 1 | 1 | 0 | 2 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 3 | 2 | 4 | 0 | 2 | 1 | 1 | 2 | 0
IMPATIENCE (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 3 | 5 | 1 | 2 | 1 | 0 | 1 | 1 | 2
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
RESTLESSNESS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 2 | 0 | 0 | 1 | 2 | 2
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.